CLINICAL TRIAL: NCT04724434
Title: Single Center Prospective Controlled Follow-up Study of COVID-19 Patients in the District Konstanz (FSC19-KN)
Brief Title: Follow-up Study of COVID-19 Patients in the District Konstanz
Acronym: FSC19-KN
Status: Completed | Type: Observational
Sponsor: Hegau-Bodensee-Klinikum Singen (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, PD Dr. med. Marc Kollum, Head of Cardiology and Internal Medicine, Hegau-Bodensee-Klinikum Singen
Other Study IDs: 20-1020
Record Dates: First submitted 2021-01-13; First posted 2021-01-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2 Positive Patients
Keywords: COVID-19 Virus disease; SARS-CoV-2; Hospitalization; Quality of life; EQ-5D-5L; Cardiomyopathy, Kansas City (KCCQ-12)
MeSH Terms: conditions — COVID-19; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In the Control group a SARS-CoV-2 antibody test will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with positive test for SARS-CoV-2 by PCR
- Control group: Patients with negative SARS-CoV-2 antibody test

SUMMARY:
This is a prospective single-center study for the follow-up of SARS-CoV-2 positive patients in the district of Konstanz (LKN). As part of the coronavirus pandemic, patients with SARS-CoV-2 infection are currently being treated in the clinics of the LKN's health network at the Singen (Hegau-Bodensee Clinic) and Konstanz (Konstanz Clinic) locations. So far, there is little data on the long-term effects of SARS-CoV-2 infection. As part of this study, the disease progression of these patients will be monitored. Study objective: Prospective, controlled follow-up observation of SARS-CoV-2 positive patients regarding their secondary diseases and quality of life.

ELIGIBILITY:
Inclusion Criteria:

A Inclusion Criteria of SARS-CoV-2 positive patients:

Patient must meet all of the following criteria.

1. Positive test for SARS-CoV-2 by PCR
2. Signed informed consent and privacy policy

B Inclusion Criteria of the control Group:

Volunteer must meet all of the following criteria.

1. No contact to SARS-CoV-2 positive patients
2. negative SARS-CoV-2 antibody test
3. Signed informed consent and privacy policy

Exclusion Criteria:

Patient/Volunteer will be excluded if any of the following conditions apply:

1. Patient/Volunteer age < 18 years
2. Patient/Volunteer who are unable to read the information and understand the nature of the study
3. Patient/Volunteer participate in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The SARS-CoV-2 positive patients in the Konstanz district are invited to participate in the study by information letter. The addressing and sending of the study documents will take place via the Health Department of the district of Konstanz. The study team only gets knowledge of those positively tested patients who responded to the cover letter and declare their informed consent to the study.
  Probands for the control group will be contacted and invited to the study by announcements in local newspapers and flyers in our hospital. Only those probands are included to the study, who can be matched to one participant of the SARS-CoV-2 positive group by age, gender and cardiovascular risk factors such as smoking, diabetes mellitus and arterial hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Hospitalization | Between 1 year after enrollment and 5 years after last patient in
  Primary endpoint

SECONDARY OUTCOMES:
EQ-5D-5L | Between 1 year after enrollment and 5 years after last patient in
  Secondary endpoint
KCCQ-12 | Between 1 year after enrollment and 5 years after last patient in
  Secondary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kollum, PD Dr. med., Principal Investigator — Hegau-Bodensee-Klinikum Singen
Locations (1):
- Hegau-Bodensee-Klinikum Singen, Singen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haberland E, Haberland J, Richter S, Schmid M, Hromek J, Zimmermann H, Geng S, Winterer H, Schneider S, Kollum M. Seven Months after Mild COVID-19: A Single-Centre Controlled Follow-Up Study in the District of Constance (FSC19-KN). Int J Clin Pract. 2022 Aug 12;2022:8373697. doi: 10.1155/2022/8373697. eCollection 2022. PMID 36035510
- [Background] Kohler AK, Richter S, Schmid M, Zimmermann H, Winterer H, Schneider S, Kollum M. Three-Year Follow-Up of COVID-19 Cases in District of Constance, Germany. A Prospective, Controlled Cohort Study (FSC19-KN). J Clin Med. 2025 Feb 21;14(5):1439. doi: 10.3390/jcm14051439. PMID 40094912